CLINICAL TRIAL: NCT00355771
Title: Placebo Controlled Pilot Study on the Efficacy of Levocetirizine 5 mg in Reducing Symptoms, Airway Resistance, and Sleep Impairment in Patients With Persistent Allergic Rhinitis
Brief Title: Levocetirizine 5 mg: Reduction of Symptoms, Airway Resistance and Sleep Impairment in Persistent Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut für Atemwegsforschung GmbH (Industry)
Collaborators: UCB Pharma (Industry)
Responsible Party: Claus Bachert, MD PhD, Institut für Atemwegsforschung GmbH
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-1-2005
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis; histamine antagonist; sleep disorder
MeSH Terms: conditions — Rhinitis, Allergic; Sleep Wake Disorders | interventions — levocetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group 1 (Experimental)
  Interventions: Drug: Levocetirizine
- Treatment Group 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levocetirizine — Intake of 1 tablet of Levocetirizine 5mg OD for 8 weeks
  Arms: Treatment Group 1
Drug: Placebo — 1 tablet OD in the morning for 8 weeks
  Arms: Treatment Group 2

SUMMARY:
The purpose of this study is to investigate, whether levocetirizine 5 mg relieves nasal and ocular symptoms of persistent allergic rhinitis and reduces increased airway resistance and sleep impairment due to this condition.

DETAILED DESCRIPTION:
Levocetirizine 5 mg is well established as the treatment of seasonal and perennial rhinoconjunctivitis. This study has been designed, to investigate its efficacy in patients suffering from persistent allergic rhinitis as defined by the ARIA (Allergic Rhinitis and its Impact on Asthma) working group of the WHO.

The study is divided in an 8 ± 2 day screening and a 56 ± 3 day treatment phase. During both periods patients keep a diary reporting on the severity of their nasal and ocular complaints, the use of rescue medication (cromoglycate eye drops and nasal spray), other concomitant medication and adverse events. They apply a 0 to 3 point score (0 = no, 1= mild, 2 = moderate, 3 = severe symptoms) to rate nasal obstruction, rhinorrhea, nasal itching, sneezing and ocular symptoms in regard to their experience during the preceding 24 hours. During the treatment period they additionally report the time of intake of study medication and their assessments of their nasal peak inspiratory flow (NPIF). NPIF is measured every evening before symptom scoring and additionally before each intake of rescue nasal spray. A device similar to the peak flow meters employed for monitoring bronchial asthma is used. Before the treatment period in its middle and at its end patients undergo a polysomnography. Furthermore 2 weeks after the start of treatment and at its end patients and investigators employ a 5-step scale (1 = very good, 2 = good, 3 = moderate, 4 = poor, 5= not at all effective) to assess the efficacy of the study medication.

Efficacy is to be established by comparison of a levocetirizine and a placebo treated group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who demonstrate their willingness to participate in the study and to comply with its procedures by signing a written informed consent.
* Subjects aged between 18 and 50 years (inclusively), of either sex and any race.
* Women of childbearing potential have to use an acceptable method of birth control.
* Subjects have to be able to understand and to adhere to the dosing and visit schedules, and to agree to record symptom scores, NPIF measurements, adverse events, concomitant medications and intake of rescue medication accurately and consistently in a daily diary.
* Subjects have to suffer from symptoms of allergic rhinitis on more than 4 days a week and for more than 4 weeks per year (ARIA criteria).
* History of at least two years of persistent allergic rhinitis (as defined by ARIA criteria).
* T5SS (Total Five Symptom Score, sum of scores evaluating the severity of five symptoms of rhinoconjunctivitis) assessed on visit 1 is > 8; in particular, nasal obstruction is rated ≥ 2.
* A CAP or prick test obtained within 12 months before visit 1 demonstrating sensitization to one or more allergens which anticipate symptoms of persistent allergic rhinitis on at least 4 days per week during the treatment period.
* On visit 2: Average T5SS calculated from diary reports is > 8 during the screening period; average rating of nasal obstruction is ≥ 2.

Exclusion Criteria:

* Women who are pregnant or nursing.
* Subjects who have not observed the designated washout periods for any of the prohibited medications.
* Subjects unable to understand the nature, scope, and possible consequences of the study or being suspected of non-compliance.
* Subjects who have used any investigational product within 30 days prior to enrollment or any investigational antibodies for asthma or allergic rhinitis in the past 90 days.
* History of alcohol or drug abuse.
* Any disease of the upper and lower respiratory tract except for allergic rhinitis during the last 2 weeks before visit 1, 2 and 3; any significant impairment of nasal patency.
* Subjects with current evidence of hematopoietic, cardiovascular, hepatic, renal, neurologic, psychiatric or autoimmune disease; or a tumor or conditions which may interfere with the absorption, distribution, metabolism or excretion of the study medication.
* Any deviation from normal in physical examination and any disease (except for allergic rhinoconjunctivitis), which might deteriorate significantly due to the subject's participation, or require impermissible medication or interfere with study evaluation.
* History of hypersensitivity to the study drug or its excipients.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2006-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Average T5SS calculated with respect to the 8 week treatment period. T5SS is the daily sum of 4-step symptom scores, which patients use to report the severity of five symptoms of allergic rhinoconjunctivitis in their diaries. | 8 week treatment period

SECONDARY OUTCOMES:
Average of the individual symptom scores | 8 week treatment period
average daily NPIF | 8 week treatment period
average use of rescue medication | 8 week treatment period
sleep quality parameters assessed by polysomnography | in the beginning and after 6 to 8 weeks of treatment
global valuation of the efficacy | after 4 and 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Claus Bachert, MD, PhD, Principal Investigator — Institut für Atemwegsforschung
Locations (1):
- Department of ORL, West China Hospital, Sichuan Hospital, Chengdu, Sichuan, China